CLINICAL TRIAL: NCT04269291
Title: An Investigation Into an Objective Measure of Muscle Quality, Function and Ability
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Principal Investigator, Stephanie Wentworth, Chief Investigator, Cardiff and Vale University Health Board
Other Study IDs: 7703
Record Dates: First submitted 2020-01-15; First posted 2020-02-13 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Electric Impedance; Healthy Volunteers
Keywords: electrical impedance; skeletal muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment of muscular function, quality and ability is of high importance in a diverse range of clinical disciplines from anaesthetics to physiotherapy. This study will look at the range of measurement techniques currently in use and development and considers their effectiveness and objectivity. It will also investigate whether an objective measurement technique can be found or developed that can be used both in the clinical environment and the community setting. This will focus on upper limb function and ability; ability is used here instead of strength since ability better describes functions needed for daily living rather than the maximum output a muscle is capable of.

DETAILED DESCRIPTION:
A literature review (available on request) explores what can be measured, the problems of measurement and its objectivity. The aim is to investigate whether there is a method of measuring muscle quality, function and ability that can be used objectively in the clinical environment or the community with equal ease or whether such a method can be developed.

The literature review identified electrical impedance myography (EIM) as a potentially objective technique to measure muscle quality and ability. Two hypotheses are proposed to test the objectivity:

The EIM measurement of passive and active muscle is not significantly different.

EIM measurements in younger and older adult volunteers is significantly different.

There is only one study visit for this study, so all study activities will occur on the same day at the Posture and Mobility Centre, Treforest or the Artificial Limb and Appliance Centre, Rookwood Hospital.

Eligibility for the study will be checked against the inclusion and exclusion criteria, including the requests to not have done heavy exercise for an hour before the measurements and also to have emptied their bladder before attending for the visit.

Any concerns will be also be addressed appropriately

Following the eligibility check, the CI will ensure the participant has read the PIS and fully understand it before obtaining informed consent.

Participants will be assigned a number in order to anonymise their data and only the main investigator will have access to this database of participants.

The following data will then be collected by the CI and written in a Case Report Form (CRF):

* Gender
* Date of birth (to ascertain age)
* Height (to calculate BMI)
* Weight (to calculate BMI)
* Waist measurement (to calculate RFM index, considered an alternative indicator of health).
* Medical history to ensure no existing neuromuscular, active arthritis or cardiac conditions or active implanted devices
* Perceived level of fitness - using the NHS scale https://www.nhs.uk/live-well/healthy-weight/bmi-calculator/ (to gauge muscle ability)
* A quantitative measurement method will be used in conjunction with a structured initial questionnaire relating to physical characteristics (e.g. height, weight, waist measurement, date of birth to indicate age and perceived level of fitness https://www.nhs.uk/live-well/healthy-weight/bmi-calculator/).

The CI will then attach electrodes to the arm of the participant and they will be asked to relax for 10 minutes.

The measurement device is an ImpediMed IMP SFB7 (CE 0129 marked) and is portable. EIM passes an imperceptible AC current (less than 1 mA) through the muscle under investigation and the impedance of that muscle is then recorded through a range of frequencies or at chosen frequencies.

Measurements of EIM of the relaxed muscles will be recorded in the CRF followed by measurements of EIM in the contracted muscle.

Electrodes will be carefully removed from the participant and they are invited to relax for a further 5 minutes and have a drink of water.

The participant's involvement in the study will end after the measurements have been taken.

ELIGIBILITY:
Inclusion Criteria:

* be volunteers
* be over the age of 18
* no pre-existing neuromuscular disease
* not have an implanted cardiac device
* be well at the time of measurement
* be able to give informed consent

Exclusion Criteria:

* Any existing neuromuscular disorder (eg multiple sclerosis, ALS, MND, CP)
* Any existing cardiac disease (including having a pacemaker or ICD)
* Active arthritis
* Be pregnant
* Any other implanted electrical device
* Not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Observation of healthy volunteer measurement of Electrical Impedance Myography in arm muscles. | One visit per volunteer. Data to be accumulated over approximately 1 year
  Primary Objective To measure EIM in sketetal arm muscle. Measurements to be made when the muscles are passive and when they are contracted.
  EIM measurements are reactance and resistance which are both measured in Ohms.
  At least 20 eligible and consented volunteers to be recruited and measured.
  To be measured at the one healthy volunteer visit. No other visits are part of the study.

SECONDARY OUTCOMES:
Age of participants | through study completion, an average of 1 year
  DOB recorded to classify healthy volunteers into age ranges.
  This will be recorded at the one visit.
Fitness health measure of participants | through study completion, an average of 1 year
  To calculate an indication of the health of the volunteers the following will be measured and recorded.
  Height (m) Weight (kg) waist size (cm) Measured to calculate BMI index and RFM index (considered an alternative indicator of health).
  All will be measured at the one visit. .

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wentworth, Principal Investigator — stephanie.wentworth@wales.nhs.uk
Locations (1):
- Cardiff and Vale University Health Board., Cardiff, United Kingdom